CLINICAL TRIAL: NCT07397442
Title: A Prospective, Phase II, Single-Arm Study on the Efficacy and Safety of Neoadjuvant Short-Course Radiotherapy Combined With Chemotherapy and Immunotherapy in Mid-Low Locally Advanced Rectal Cancer
Brief Title: Short-Course Radiotherapy Combined With Chemotherapy and Immunotherapy in Mid-Low Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Yingchi Yang, Professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2026-P2-013-01
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Rectal Cancer, Adenocarcinoma; Rectal Cancer Stage II; Rectal Cancer Stage III
Keywords: locally advanced rectal cancer; short-course radiotherapy; anti-PD1; anti-CTLA4; complete response
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response | interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Short-course radiotherapy plus chemo-immunotherapy (Experimental)
  Interventions: Combination Product: Short-Course Radiotherapy Combined with Chemotherapy and Immunotherapy

INTERVENTIONS:
Combination Product: Short-Course Radiotherapy Combined with Chemotherapy and Immunotherapy — ● Radiotherapy: Total dose of 25 Gy delivered in 5 fractions, 5 Gy per fraction, over a total course of 5 days (Target area: Only the gross rectal tumor and radiologically suspected metastatic positive lymph nodes, without irradiation of additional lymphatic drainage areas).
  * Qibei'an (Iparolizumab-tovorilimab Injection):
    5 mg/kg intravenous drip, administered once 2 days after radiotherapy completion.
  * Camrelizumab:
    200 mg intravenous drip, administered sequentially 3 times after Qibei'an, each in combination with XELOX chemotherapy.
  * XELOX Chemotherapy:
  Oxaliplatin 130 mg/m2 intravenous drip, Day 1; Capecitabine 1000 mg/m2 orally twice daily, Day 1 to Day 14.

SUMMARY:
The goal of this clinical trial is to test a new combination treatment for locally advanced rectal cancer (cancer in the lower or middle part of the rectum that has not spread to distant organs). The study aims to increase the chance of making the tumor disappear completely (called "complete response") and improve the quality of life by increasing the rate of anal sphincter preservation (avoiding permanent colostomy bags).

The main questions it aims to answer are:

Does the combination of short-course radiation therapy, two types of immunotherapy drugs (Qibeian and Aike), and chemotherapy (XELOX) increase the complete response rate to over 50%? Is this combination treatment safe, and what are the side effects? Can this treatment help more patients keep their anal function and avoid permanent stomas?

This is a single-arm study, meaning all participants will receive the experimental treatment (there is no placebo or control group).

Participants will:

Receive short-course radiation therapy (25 Gy total, given once daily for 5 consecutive days). The radiation will target only the tumor and visible lymph nodes, intentionally avoiding unaffected lymph node areas to protect the immune system.

Receive Qibei'an (a dual immunotherapy drug targeting both PD-1 and CTLA-4) once, 2 days after completing radiation.

Receive Camrelizumab (a PD-1 immunotherapy drug) three times, combined with XELOX chemotherapy.

Receive XELOX chemotherapy (Oxaliplatin ivgtt on Day 1, plus Capecitabine pills taken twice daily for 14 days, for each cycle) for up to 3 cycles.

Undergo detailed assessments after treatment, including MRI scans, colonoscopy with biopsies, and blood tests (including ctDNA tests), to determine if the tumor has disappeared or if surgery is needed.

Attend regular follow-up visits for up to 5 years after treatment (or surgery) to monitor for recurrence and assess quality of life.

The study will enroll approximately 19 patients at Beijing Friendship Hospital, Capital Medical University. An independent safety monitoring board will regularly review the data to ensure participant safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. ECOG performance status score 0-2.
3. Rectal adenocarcinoma confirmed by colonoscopic pathology, with pMMR or MSS.
4. Imaging studies confirm no distant metastasis or lateral lymph node metastasis; MRI staging is II/III (excluding T4b, N1c, N2) and any positive lymph nodes (if present) are confined within the mesorectum.
5. MRI shows the distal margin of the tumor is ≤10 cm from the anal verge, and the mesorectal fascia (MRF) is negative.
6. The longest diameter of the rectal cancer lesion is ≥10 mm on baseline CT or MRI (meeting the definition of a "measurable lesion" per RECIST 1.1 criteria).
7. Willing and able to comply with the study procedures.
8. Consent to the use of tissue and blood samples by the investigator for medical research purposes.
9. No prior history of radiotherapy or immunotherapy.
10. No history of immune system diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis, systemic vasculitis, scleroderma, pemphigus, dermatomyositis, mixed connective tissue disease, autoimmune hemolytic anemia, ulcerative colitis, HIV infection, etc.).
11. No history of endocrine system diseases (e.g., hyperthyroidism, hypothyroidism, thyroid nodules, thyroiditis, type 1 diabetes, type 2 diabetes, gestational diabetes, other specific types of diabetes, Cushing's syndrome, primary aldosteronism, pheochromocytoma, adrenal insufficiency, pituitary adenoma, anterior pituitary hypofunction, acromegaly, gigantism, polycystic ovary syndrome, precocious puberty, hypogonadism, hyperparathyroidism, hypoparathyroidism, etc.).
12. No severe cardiac, pulmonary, hepatic, or renal dysfunction.
13. No jaundice or gastrointestinal obstruction.
14. No concurrent acute infection.
15. Subjects must undergo all required baseline laboratory assessments, and results must be obtained within 1 week before enrollment. Laboratory values must meet the following criteria (per CTCAE 5.0):

    1. White blood cell count ≥2000/μL.
    2. Neutrophil count ≥1500/μL.
    3. Platelet count ≥100×10³/μL.
    4. Hemoglobin ≥9.0 g/dL.
    5. Creatinine: serum creatinine ≤1.5 × upper limit of normal (ULN) or creatinine clearance >50 mL/min (calculated using the Cockcroft-Gault formula).
    6. Creatinine clearance for females = [140 - age (years)] × weight (kg) × 0.85 ÷ [72 × serum creatinine (mg/dL)].
    7. Creatinine clearance for males = [140 - age (years)] × weight (kg) × 1.00 ÷ [72 × serum creatinine (mg/dL)].
    8. Aspartate aminotransferase (AST) ≤3 × ULN, alanine aminotransferase (ALT) ≤3 × ULN, total bilirubin ≤1.5 × ULN.
16. No psychiatric/psychological disorders affecting social functioning.
17. Women of childbearing potential must have a negative serum pregnancy test (blood HCG) within 1 week before enrollment.
18. Women of childbearing potential and men who are sexually active with women of childbearing potential must agree to use appropriate contraceptive methods.

Exclusion Criteria:

1. Multifocal cancer, or concomitant other malignant tumors.
2. Received any anti-tumor therapy for other malignant tumors within the past 5 years.
3. Underwent major surgery recently (within 6 months).
4. Presence of multiple factors affecting oral drug absorption (e.g., inability to swallow, nausea, vomiting, chronic diarrhea, intestinal obstruction, etc.).
5. Any uncontrolled, severe comorbid diseases.
6. Allergy to any component of the study medication.
7. Life expectancy less than 5 years for any reason.
8. Planning to undergo or previously underwent organ/bone marrow transplantation.
9. Received immunosuppressive agents or glucocorticoid therapy aimed at suppressing immune responses within 1 month before enrollment.
10. For patients with a history of central nervous system diseases, the investigator will determine whether their current condition allows them to provide informed consent or comply with the study procedures, and subsequently decide whether they can be enrolled.
11. Other diseases or conditions that may prevent completion of the study treatment (e.g., alcoholism, drug addiction, etc.).
12. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2033-02-28 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | Approximately 4 months after treatment starts
  Including both clinical and pathological complete response

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang Y, Pang K, Lin G, Liu X, Gao J, Zhou J, Xu L, Gao Z, Wu Y, Li A, Han J, Wu G, Wang X, Li F, Ye Y, Zhang J, Chen G, Wang H, Kong Y, Wu A, Xiao Y, Yao H, Zhang Z. Neoadjuvant chemoradiation with or without PD-1 blockade in locally advanced rectal cancer: a randomized phase 2 trial. Nat Med. 2025 Feb;31(2):449-456. doi: 10.1038/s41591-024-03360-5. Epub 2025 Jan 6. PMID 39762418